CLINICAL TRIAL: NCT01702298
Title: An Open-label Study to Assess the Safety and Tolerability of MK-0431D for the Treatment of Patients With Type 2 Diabetes Mellitus (T2DM) With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: A Study to Assess the Safety and Tolerability of Sitagliptin/Simvastatin Fixed-dose Combination (FDC) in Participants With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Metformin Monotherapy (MK-0431D-312)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0431D-312
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Simvastatin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitagliptin 100 mg/simvastatin 40 mg FDC (Experimental): Sitagliptin 100 mg/simvastatin 40 mg FDC once daily in the evening for 6 weeks. Participants will continue pre-study dose of metformin >=1000 mg per day.
  Interventions: Drug: Sitagliptin 100 mg/simvastatin 40 mg FDC; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin 100 mg/simvastatin 40 mg FDC — Sitagliptin 100 mg/simvastatin 40 mg FDC tablet administered once daily in the evening for 6 weeks
  Other Names: MK-0431D
Drug: Metformin — Participants will continue pre-study dose of metformin tablet(s) >=1000 per day
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®; Metgluco®; Glycoran®

SUMMARY:
The purpose of this study is to examine the safety and tolerability of sitagliptin 100 mg/simvastatin 40 mg FDC (MK-0431D) in Vietnamese participants with type 2 diabetes mellitus with inadequate glycemic control on metformin.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Male, or female who is not of reproductive potential or if of reproductive potential agrees to abstain or use (or have their partner use) two acceptable methods of birth control during the study and for 14 days after the last dose of study drug
* Currently on metformin monotherapy (>=1000 mg per day) for at least 4 weeks prior to study participation
* Not on statin therapy or other lipid-lowering agent for at least 6 weeks prior to study participation

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of 2 or more episodes of hypoglycemia resulting in seizure, coma or loss of consciousness over the past 3 months
* On a thiazolidinedione (TZD) within the past 12 weeks
* Has been treated with a statin or other lipid-lowering agent within 6 weeks prior to study participation
* Is on or likely to require treatment with a prohibited medication (itraconazole, ketoconazole, posaconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, nefazodone, gemfibrozil, cyclosporine, danazol, amiodarone, verapamil, diltiazem, amlodipine, ranolazine, niacin)
* Intends to consume >1.2 liters of grapefruit juice per day during the study
* Is on or likely to require treatment for >=2 consecutive weeks or repeated courses of corticosteroids (inhaled, nasal and topical corticosteroids are permitted)
* Is on a weight loss program and not in the maintenance phase or has started a weight loss medication or has undergone bariatric surgery within 12 months prior to study participation
* Has undergone a surgical procedure within 4 weeks of study participation or has planned major surgery during the study
* History of myopathy or rhabdomyolysis with any statin
* History of myocardial infarction, unstable or stable angina, angioplasty, bypass surgery, myocardial ischemia, peripheral artery disease, abdominal aortic aneurysm, transient ischemic attacks, stroke of carotid origin or >50% obstruction of a carotid artery
* Diagnosis of congestive heart failure with New York Heart Association (NYHA) Class III or IV cardiac status
* History of active liver disease (other than non-alcoholic steatosis) including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Chronic progressive neuromuscular disorder
* Human immunodeficiency virus (HIV)
* Hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Currently being treated for hyperthyroidism or is on thyroid hormone replacement therapy and has not been on a stable dose for at least 6 weeks
* History of malignancy <=5 years prior to study participation, except for basal cell or squamous cell skin cancer or in situ cervical cancer
* Positive urine pregnancy test
* Pregnant or breastfeeding, or is expecting to conceive or donate eggs during the study, including 14 days following the last dose of study drug
* User of recreational or illicit drugs or has had a recent history of drug abuse
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2013-05-29 (Actual); Study Completion 2013-05-29 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431D-312&kw=0431D-312&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin 100 mg/Simvastatin 40 mg FDC: Sitagliptin 100 mg/simvastatin 40 mg FDC once daily in the evening for 6 weeks. Participants continued on their pre-study dose of metformin (>=1000 mg per day).
Period: Overall Study
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Started | 42
Completed | 41
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 23
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 159.3 (40.9)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 109.6 (27.2)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: md/dL] | 195.2 (36.4)
(Non-High-Density Lipoprotein Cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 152.0 (37.9)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 225.3 (152.5)
High-Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 43.1 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG at Week 6 based on longitudinal data analysis (LDA) model including both baseline and post-baseline measurements as response variable and term time.
Time Frame: Baseline and Week 6
Population: Full analysis set (FAS) defined as all participants who took at least one dose of study medication and had at least one baseline or post-baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 42
mg/dL | -27.6 (58.4) [-46.0 to -9.3]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Description: An adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product.
Time Frame: Up to 8 weeks (including 14 days after final dose of study drug)
Population: All participants treated population defined as all enrolled participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 42
Percentage of participants | 9.5 [2.7 to 22.6]

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: Participants who were discontinued from study drug due to an adverse event during the 6 weeks of treatment.
Time Frame: Up to 6 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 42
Participants | 0

4. Secondary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Change from baseline in LDL-C was measured as a percent change from baseline at Week 6 based on LDA model including percent change from baseline as response variable and term time.
Time Frame: Baseline and Week 6
Population: FAS defined as all participants who took at least one dose of study medication and had both baseline and post-baseline measurements. One participant, who had no on-treatment data, was excluded from the FAS for the LDA analysis of LDL-C.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 41
Percent change | -46.5 (17.0) [-51.9 to -41.2]

5. Secondary Outcome: Change From Baseline in Total Cholesterol (TC)
Description: Change from baseline in TC was measured as a percent change from baseline at Week 6 based on LDA model including percent change from baseline as response variable and term time.
Time Frame: Baseline and Week 6
Population: FAS defined as all participants who took at least one dose of study medication and had both baseline and post-baseline measurements.
  One participant, who had no on-treatment data, was excluded from the FAS for the LDA analysis of TC.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 41
Percent change | -33.7 [-37.3 to -30.0]

6. Secondary Outcome: Change From Baseline in Non-high Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Change from baseline in non-HDL-C was measured as a percent change from baseline at Week 6 based on LDA model including percent change from baseline as response variable and term time.
Time Frame: Baseline and Week 6
Population: FAS defined as all participants who took at least one dose of study medication and had both baseline and post-baseline measurements. One participant, who had no on-treatment data, was excluded from the FAS for the LDA analysis of non-HDL-C.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 41
Percent change | -43.1 [-47.4 to -38.9]

7. Secondary Outcome: Change From Baseline in Triglycerides (TG)
Description: Change from baseline in TG was measured as a percent change from baseline at Week 6 (median and distribution free 95% confidence interval).
Time Frame: Baseline and Week 6
Population: FAS defined as all participants who took at least one dose of study medication and had both baseline and post-baseline measurements. One participant, who had no on-treatment data, was excluded from the FAS.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 41
Percent change | -31.8 (26.3) [-41.1 to -18.3]

8. Secondary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: Change from baseline in HDL-C was measured as a percent change from baseline at Week 6 based on LDA model including percent change from baseline as response variable and term time.
Time Frame: Baseline and Week 6
Population: FAS defined as all participants who took at least one dose of study medication and had both baseline and post-baseline measurements. One participant, who had no on-treatment data, was excluded from the FAS for the LDA analysis of HDL-C.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Number analyzed (Participants) | 41
Percent change | 1.3 [-5.0 to 7.5]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Arm/Group | Sitagliptin 100 mg/Simvastatin 40 mg FDC
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 3/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg/Simvastatin 40 mg FDC (N=42)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.